CLINICAL TRIAL: NCT02065050
Title: Comprehensive Intervention to Evaluate Outcomes AND Cost in Hospitalized Surgical Patients With DM: COACH-DM
Brief Title: Comprehensive Intervention to Evaluate Outcomes AND Cost in Hospitalized Surgical Patients With Diabetes Mellitus (DM)
Acronym: COACH-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Rajesh K. Garg, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012P002461; UD7HP25059 (Other Grant/Funding Number: HRSA)
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Diabetes
Keywords: Diabetes mellitus; Team approach
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Individuals in the usual care arm will not receive frequent contact by the study team. Individuals will be seen by a study team clinician 1 year after discharge to review diabetes management and obtain pertinent study related data.
- Continued care (Experimental): team-based care: Individuals in the continued care arm will be frequently contacted by the study team (consisting of endocrinologists, nurse practitioners, and health coaches) over the course of one year post-discharge. The team will monitor blood sugars and other health data, altering management as needed.
  Interventions: Other: team-based care

INTERVENTIONS:
Other: team-based care — Patients in the eDMS arm are called at least every month for their diabetes treatment.
  Arms: Continued care

SUMMARY:
This study is being performed to evaluate whether a comprehensive discharge planning and close follow up for one year can improve clinical outcomes and cut costs of care for patients with poorly controlled diabetes. The study takes a high risk approach and is focused on patients admitted to hospital for elective surgery with HbA1c >8%. Secondary goals include improving teamwork and communication for clinicians within the team and teaching nurse practitioners and physicians-in-training how to work effectively within interdisciplinary teams. Investigators anticipate that the results of this project may lead to the following benefits: 1) improved health outcomes for surgical patients with diabetes, 2) improved strategies for better communication within interdisciplinary health care teams, and 3) decreased health care costs.

DETAILED DESCRIPTION:
All patients who are planned for elective surgery at the hospital are seen in the pre-operative center a few days before admission. The diabetes management team becomes involved in care of patients with HbA1c >8.0% at this time. Once the patients are admitted to the hospital, the diabetes management team continues to follow them until they are ready for discharge. At the point of discharge, patients are randomized to one of two arms- the usual care group and the expanded diabetes management service (eDMS). The eDMS group is followed closely for 1 year after discharge by the investigators to make sure they receive appropriate care for their diabetes.

Aims of this study are:

1. To evaluate whether patients that receive the eDMS have lower re-hospitalization rates at 1 month compared to patients who receive the traditional (current) DMS. Investigators hypothesize that the eDMS program will have lower re-hospitalization rates at 1 month.
2. To evaluate whether patients that receive the eDMS have lower HbA1c levels at 1 year compared with patients who receive the traditional DMS. Investigators hypothesize that patients in the eDMS program will have lower HbA1c levels and improved diabetes-related health outcomes after 1 year in the program.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery
* HbA1c >=8% within 3 months before surgery
* Age > 18 years

Exclusion Criteria:

* undergoing same day surgery without post-operative admission
* HbA1c < 8%
* individuals undergoing bariatric surgery
* individuals with metastatic cancer or short life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 1 year after date of discharge
  Data on participant HbA1c will be collected at the end of the 1 year.

SECONDARY OUTCOMES:
Blood Pressure | 1 year after discharge
  Blood pressure measurements will be obtained at 1 year.
LDL Cholesterol | 1 year post-discharge
  LDL cholesterol measured at 1 year after discharge.
Urine microalbumin | 1 year post-discharge
  Urine microalbumin measured at 1 year after discharge.
BMI | 1-year post-discahrge
  BMI will be obtained at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh K. Garg, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
This study will not produce data that can be shared

REFERENCES:
- [Derived] Garg R, Hurwitz S, Rein R, Schuman B, Underwood P, Bhandari S. Effect of follow-up by a hospital diabetes care team on diabetes control at one year after discharge from the hospital. Diabetes Res Clin Pract. 2017 Nov;133:78-84. doi: 10.1016/j.diabres.2017.08.014. Epub 2017 Aug 24. PMID 28898714